CLINICAL TRIAL: NCT02338362
Title: The Effect of Inhaled Corticosteroids on Intraocular Pressure in Patients With Ocular Hypertension or Controlled Glaucoma.
Brief Title: Inhaled Corticosteroids: Effect on Intraocular Pressure in Patients With Controlled Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Graham E Trope, Toronto Western Hospital Glaucoma Service Co-Director, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 13-6069-A
Record Dates: First submitted 2014-12-02; First posted 2015-01-14 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Ocular Hypertension; Glaucoma, Open-Angle
Keywords: Corticosteroids; Bronchodilator Agents; Intraocular Pressure
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone (Active Comparator): 10 participants will be asked to use fluticasone propionate 250 µg metered-dose inhaler 1 puff twice-daily for 6 weeks.
  Interventions: Drug: Fluticasone propionate inhaler
- Saline placebo (Placebo Comparator): 10 participants will be asked to use a saline placebo metered-dose inhaler 1 puff twice-daily for 6 weeks.
  Interventions: Drug: Saline placebo inhaler

INTERVENTIONS:
Drug: Fluticasone propionate inhaler — fluticasone propionate 250 µg metered-dose inhaler
  Arms: Fluticasone
Drug: Saline placebo inhaler — saline metered dose inhaler
  Arms: Saline placebo

SUMMARY:
The purpose of this study is to determine whether a commonly prescribed orally inhaled corticosteroid treatment will induce a clinically meaningful elevation in intraocular pressure, when administered to patients with ocular hypertension (OHT) or open-angle glaucoma (OAG). Based on the response to high-dose corticosteroids, this patient group is more likely than the normal population to demonstrate this adverse effect.

DETAILED DESCRIPTION:
Systemic and topical ophthalmic steroids have long been associated with ocular effects, such as glaucoma or cataracts.[Alfano JE; Bernstein HN et al. 1962; Bernstein HN et al. 1963; Becker B and Mills DW in Arch Ophthalm 1963; Becker B and Mills DW in JAMA 1963; Armaly MF 1963 (1); Armaly MF 1963 (2); and Buckley RJ] Periocular steroid injections [Herschler J; Kalina RE] and steroids applied to periocular skin [Aggarwal RK et al.] have also been reported to increase intraocular pressure (IOP) and raised IOP is the major risk factor for glaucoma.

Ocular hypertension (OHT) is defined as an IOP above 21mmHg in one or both eyes without detectable glaucomatous damage. Primary open-angle glaucoma (POAG) is a chronic and progressive optic neuropathy of unknown etiology characterized by disc cupping, and often associated with visual field defects and elevated IOP. This disease is one of the leading causes of blindness worldwide.[Kwon YH et al.] Approximately 18% to 36% of the general population are corticosteroid responders. This response is increased to 46% to 92% in patients with POAG.[Tripathi RC et al.] Asthma is the most common chronic respiratory illness in Canada, affecting approximately 10% of the population. For the majority of these patients, long-term inhaled corticosteroids (ICS) are standard of care to prevent acute asthma exacerbations.[Kim H and Mazza J] Although the systemic absorption of inhaled and nasal steroids has been established, the clinically relevant ocular side effects are poorly defined. [Cave A et al.; Allen DB et al.] A large prospective study in 1995 by Samiy et al reported no statistically significant increase of IOP in 187 patients without glaucoma taking inhaled steroids for various pulmonary conditions.[Samiy N et al.] However, six cases of increased IOP associated with combined nasal and inhaled steroid use in non-glaucomatous patients have been reported. [Dreyer EB; Desnoeck M et al.; Opatowsky I et al.] A large case-control study in 1997 suggested that current users of high doses of ICS prescribed regularly for 3 or more months were at increased risk of OHT or OAG (OR 1.44; 95% CI 1.01-2.06).[Garbe E et al.] In contrast, Gozalez et al. conducted a nested case-control study in 2010 with Quebec data which showed current and continuous use of ICS did not result in increased risk of glaucoma or raised IOP requiring treatment.[Gonzalez AV et al.] Similarly, Duh et al. reported no association between inhaled budesonide daily therapy and increased IOP in 1255 asthmatic patients.[Duh MS et al.] Further, a prospective population-based cohort study published in 2012 suggested no association between the development of OAG and ICS in the elderly.[Marcus MW et al.] In 2013, our group published a randomized double-masked controlled trial that showed no evidence of IOP elevation after 6 weeks use of beclomethasone nasal spray in 19 patients with OHT and POAG.[Yuen D et al.] The purpose of the current study protocol would be to extend the study to investigate ICS in the same patient population.

To date, the effect of inhaled corticosteroids in those with pre-existing OHT or POAG remains uncertain. Considering the large number of patients on inhaled steroids, investigating the use of inhaled steroid in glaucoma patients could have significant clinical impact. This study was designed to evaluate the effect of inhaled fluticasone propionate on intraocular pressure (IOP) in patients with OHT or controlled open-angle glaucoma (OAG).

Patient randomization was performed by an independent Research Coordinator in a separate physical space and kept sealed from the principal study investigators, who assessed and recorded outcome measures, until the completion of study data collection. IOP was measured in a masked fashion, using a second observer to record values. Two measurements within 1 mmHg were averaged for each data point. With a sample size of 8 patients per interventional arm, the study is powered at 0.80 to detect an elevation of 3.2 mmHg (≥20%) from mean, assuming a standard deviation of 2.5 mmHg. Baseline data will be compared between groups using the student's t test and Fisher exact test. A 2-sided p value of <0.05 will be considered statistically significant. The primary outcome measure (mean IOP) will be assessed using a 1-sided Student t test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years, inclusive
* Mild-moderate open-angle glaucoma/ocular hypertension with cup:disc ratio <0.85 vertically and humphrey visual field mean deviation >-12.00 (BOTH EYES must meet this criteria for patient to be included)
* Glaucoma well-controlled, defined by IOP < 21 mmHg and at target with no visual field/disc progression for at least 6 months (BOTH EYES must meet this criteria for patient to be included)

Exclusion Criteria:

* Any form of steroid medication use within the prior 6 weeks
* Any previous intra-ocular surgery or refractive surgery in the study eye
* no light perception (i.e. blindness) in either eye
* unwilling/unable to give consent
* unwilling to accept randomization
* patient potentially unavailable for follow-up visits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham E Trope, MD,PhD,FRCSC, Principal Investigator — University Health Network, Toronto Western Hospital

REFERENCES:
- [Background] ALFANO JE. CHANGES IN THE INTRAOCULAR PRESSURE ASSOCIATED WITH SYSTEMIC STEROID THERAPY. Am J Ophthalmol. 1963 Aug;56:245-7. doi: 10.1016/0002-9394(63)91858-0. No abstract available. PMID 14061602
- [Background] BERNSTEIN HN, SCHWARTZ B. Effects of long-term systemic steroids on ocular pressure and tonographic values. Arch Ophthalmol. 1962 Dec;68:742-53. doi: 10.1001/archopht.1962.00960030746009. No abstract available. PMID 13967694
- [Background] BERNSTEIN HN, MILLS DW, BECKER B. Steroid-induced elevation of intraocular pressure. Arch Ophthalmol. 1963 Jul;70:15-8. doi: 10.1001/archopht.1963.00960050017005. No abstract available. PMID 13967695
- [Background] BECKER B, MILLS DW. CORTICOSTEROIDS AND INTRAOCULAR PRESSURE. Arch Ophthalmol. 1963 Oct;70:500-7. doi: 10.1001/archopht.1963.00960050502012. No abstract available. PMID 14078872
- [Background] BECKER B, MILLS DW. ELEVATED INTRAOCULAR PRESSURE FOLLOWING CORTICOSTEROID EYE DROPS. JAMA. 1963 Sep 14;185:884-6. doi: 10.1001/jama.1963.03060110088027. No abstract available. PMID 14043096
- [Background] ARMALY MF. EFFECT OF CORTICOSTEROIDS ON INTRAOCULAR PRESSURE AND FLUID DYNAMICS. I. THE EFFECT OF DEXAMETHASONE IN THE NORMAL EYE. Arch Ophthalmol. 1963 Oct;70:482-91. doi: 10.1001/archopht.1963.00960050484010. No abstract available. PMID 14078870
- [Background] ARMALY MF. EFFECT OF CORTICOSTEROIDS ON INTRAOCULAR PRESSURE AND FLUID DYNAMICS. II. THE EFFECT OF DEXAMETHASONE IN THE GLAUCOMATOUS EYE. Arch Ophthalmol. 1963 Oct;70:492-9. doi: 10.1001/archopht.1963.00960050494011. No abstract available. PMID 14078871
- [Background] Buckley RJ. Allergic eye disease--a clinical challenge. Clin Exp Allergy. 1998 Dec;28 Suppl 6:39-43. doi: 10.1046/j.1365-2222.1998.0280s6039.x. PMID 9988434
- [Background] Herschler J. Intractable intraocular hypertension induced by repository triamcinolone acetonide. Am J Ophthalmol. 1972 Sep;74(3):501-4. doi: 10.1016/0002-9394(72)90916-6. No abstract available. PMID 5053696
- [Background] Kalina RE. Increased intraocular pressure following subconjunctival corticosteroid administration. Arch Ophthalmol. 1969 Jun;81(6):788-90. doi: 10.1001/archopht.1969.00990010790006. No abstract available. PMID 5783749
- [Background] Aggarwal RK, Potamitis T, Chong NH, Guarro M, Shah P, Kheterpal S. Extensive visual loss with topical facial steroids. Eye (Lond). 1993;7 ( Pt 5):664-6. doi: 10.1038/eye.1993.152. PMID 8287990
- [Background] Kwon YH, Fingert JH, Kuehn MH, Alward WL. Primary open-angle glaucoma. N Engl J Med. 2009 Mar 12;360(11):1113-24. doi: 10.1056/NEJMra0804630. No abstract available. PMID 19279343
- [Background] Tripathi RC, Parapuram SK, Tripathi BJ, Zhong Y, Chalam KV. Corticosteroids and glaucoma risk. Drugs Aging. 1999 Dec;15(6):439-50. doi: 10.2165/00002512-199915060-00004. PMID 10641955
- [Background] Kim H, Mazza J. Asthma. Allergy Asthma Clin Immunol. 2011 Nov 10;7 Suppl 1(Suppl 1):S2. doi: 10.1186/1710-1492-7-S1-S2. PMID 22165976
- [Background] Cave A, Arlett P, Lee E. Inhaled and nasal corticosteroids: factors affecting the risks of systemic adverse effects. Pharmacol Ther. 1999 Sep;83(3):153-79. doi: 10.1016/s0163-7258(99)00019-4. PMID 10576291
- [Background] Allen DB, Bielory L, Derendorf H, Dluhy R, Colice GL, Szefler SJ. Inhaled corticosteroids: past lessons and future issues. J Allergy Clin Immunol. 2003 Sep;112(3 Suppl):S1-40. doi: 10.1016/s0091-6749(03)01859-1. PMID 14515117
- [Background] Samiy N, Walton DS, Dreyer EB. Inhaled steroids: effect on intraocular pressure in patients without glaucoma. Can J Ophthalmol. 1996 Apr;31(3):120-3. PMID 8743219
- [Background] Dreyer EB. Inhaled steroid use and glaucoma. N Engl J Med. 1993 Dec 9;329(24):1822. doi: 10.1056/nejm199312093292420. No abstract available. PMID 8232507
- [Background] Desnoeck M, Casteels I, Casteels K. Intraocular pressure elevation in a child due to the use of inhalation steroids--a case report. Bull Soc Belge Ophtalmol. 2001;(280):97-100. PMID 11486469
- [Background] Opatowsky I, Feldman RM, Gross R, Feldman ST. Intraocular pressure elevation associated with inhalation and nasal corticosteroids. Ophthalmology. 1995 Feb;102(2):177-9. doi: 10.1016/s0161-6420(95)31039-1. PMID 7862403
- [Background] Garbe E, LeLorier J, Boivin JF, Suissa S. Inhaled and nasal glucocorticoids and the risks of ocular hypertension or open-angle glaucoma. JAMA. 1997 Mar 5;277(9):722-7. PMID 9042844
- [Background] Gonzalez AV, Li G, Suissa S, Ernst P. Risk of glaucoma in elderly patients treated with inhaled corticosteroids for chronic airflow obstruction. Pulm Pharmacol Ther. 2010 Apr;23(2):65-70. doi: 10.1016/j.pupt.2009.10.014. Epub 2009 Nov 1. PMID 19887116
- [Background] Duh MS, Walker AM, Lindmark B, Laties AM. Association between intraocular pressure and budesonide inhalation therapy in asthmatic patients. Ann Allergy Asthma Immunol. 2000 Nov;85(5):356-61. doi: 10.1016/S1081-1206(10)62545-8. PMID 11101175
- [Background] Marcus MW, Muskens RP, Ramdas WD, Wolfs RC, De Jong PT, Vingerling JR, Hofman A, Stricker BH, Jansonius NM. Corticosteroids and open-angle glaucoma in the elderly: a population-based cohort study. Drugs Aging. 2012 Dec;29(12):963-70. doi: 10.1007/s40266-012-0029-9. PMID 23150239
- [Background] Yuen D, Buys YM, Jin YP, Alasbali T, Trope GE. Effect of beclomethasone nasal spray on intraocular pressure in ocular hypertension or controlled glaucoma. J Glaucoma. 2013 Feb;22(2):84-7. doi: 10.1097/IJG.0b013e3182254811. PMID 21716127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,960 records of glaucoma patients with scheduled visits in a university-based glaucoma clinic were screened between August 1, 2014 and November 7, 2014.
Pre-assignment Details: 22 consented to participate and 20 completed the study.
Groups:
- Steroid Inhaler: randomized to 6 weeks of 1 puff twice daily 250ug fluticasone propionate inhaled.
- Placebo Inhaler: randomized to 6 weeks of 1 puff twice daily saline inhaled.
Period: Overall Study
Arm/Group | Steroid Inhaler | Placebo Inhaler
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone: participants will be asked to use fluticasone propionate 250 µg metered-dose inhaler 1 puff twice-daily for 6 weeks.
- Saline Placebo: participants will be asked to use a saline placebo metered-dose inhaler 1 puff twice-daily for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Fluticasone | Saline Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.0) | 65.7 (11.0) | 65.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20
Mean intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 14.3 (3.0) | 15.6 (3.6) | 15.0 (3.3)
Mean number of ocular hypotensive medications [Mean (Standard Deviation); unit: medication classes] | 1.3 (0.7) | 1.3 (1.4) | 1.3 (1.0)
Prior laser trabeculoplasty [Number; unit: participants] | 1 | 0 | 1
Mean central corneal thickness [Mean (Standard Deviation); unit: micrometers] | 553.1 (31.7) | 549.1 (30.8) | 551.1 (31.25)
Mean cup-disc ratio [Mean (Standard Deviation); unit: cup:disc ratio] — The cup-to-disc ratio compares the diameter of the cup portion of the optic disc with the total diameter of the optic disc. A cup-to-disc ratio > 0.5 might be indicative of glaucoma.
  cup:disc ratio | 0.49 (0.2) | 0.38 (0.2) | 0.44 (0.2)
Mean visual field mean deviation [Mean (Standard Deviation); unit: decibels (dB)] | -0.72 (2.6) | -1.13 (2.5) | -0.92 (2.6)
Mean logMAR visual acuity [Mean (Standard Deviation); unit: logMAR] — 20/20 vision corresponds with a logMAR score of 0, while negative logMAR scores indicate better than 20/20 vision, values > 0.5 correspond with low vision, and values > 1.3 correspond with blindness.
  logMAR | 0.19 (0.1) | 0.18 (0.1) | 0.18 (0.1)
Diagnosis [Number; unit: participants]
  Ocular Hypertension | 1 | 4 | 5
  Primary Open-Angle Glaucoma | 6 | 4 | 10
  Pigment Dispersion Glaucoma | 3 | 1 | 4
  Pseudoexfoliative Glaucoma | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure
Description: Masked assessment of intraocular pressure using goldmann application tonometry. Mean of 2 measurements within 1 mmHg will be recorded.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fluticasone | Saline Placebo
Number analyzed (Participants) | 10 | 10
mmHg | 14.7 (2.4) | 14.8 (3.8)

2. Secondary Outcome: Mean Visual Acuity
Description: best corrected logMAR visual acuity for each eye. 20/20 vision corresponds with a logMAR score of 0, while negative logMAR scores indicate better than 20/20 vision, values > 0.5 correspond with low vision, and values > 1.3 correspond with blindness.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Fluticasone | Saline Placebo
Number analyzed (Participants) | 10 | 10
logMAR | 0.15 (0.12) | 0.15 (0.08)

3. Secondary Outcome: Side Effects
Description: subjective (reported) and objective (slit lamp examination) side-effects attributable to study medications
Time Frame: from baseline to week 6
Measure: Number; unit: participants
Arm/Group | Fluticasone | Saline Placebo
Number analyzed (Participants) | 10 | 10
participants
  lens opacity | 0 | 0
  throat discomfort | 1 | 1
  headache | 1 | 0
  difficulty sleeping | 0 | 1
  no adverse effects | 8 | 8

4. Secondary Outcome: Intraocular Pressure Elevation >20% From Baseline
Description: Participants with 2 consecutive intraocular pressure measurements exceeding 20% increase from baseline were discontinued from study.
Time Frame: within 6-week observation period
Measure: Number; unit: participants
Arm/Group | Fluticasone | Saline Placebo
Number analyzed (Participants) | 10 | 10
participants
  elevation >20% | 1 | 0
  no elevation >20% | 9 | 10

5. Secondary Outcome: Adherence
Description: Adherence was calculated from self-reported study diaries and correlated to a counter that measured number of inhaled puffs built into the placebo metered-dose inhalers
Time Frame: Completion of study, up to 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of required doses
Arm/Group | Fluticasone | Saline Placebo
Number analyzed (Participants) | 10 | 10
percentage of required doses | 93.6 (7.1) | 96.1 (4.4)

ADVERSE EVENTS:
Time Frame: 6 weeks of study
Description: Patients were asked about any side-effects they were experiencing at each biweekly study visit.
Arm/Group | Fluticasone | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone (N=10) | Saline Placebo (N=10)
sore throat (General disorders) | 1 (1) | 1 (1)
headache (General disorders) | 1 (1) | 0 (0)
difficulty sleeping (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No